CLINICAL TRIAL: NCT06154447
Title: A Phase 1, Study of VX-828 in Healthy Subjects and in Subjects With Cystic Fibrosis
Brief Title: Evaluation of VX-828 in Healthy Participants and in Participants With Cystic Fibrosis
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Vertex Pharmaceuticals Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VX23-828-001
Record Dates: First submitted 2023-11-23; First posted 2023-12-04 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2025-09

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis | interventions — Itraconazole; Midazolam; tezacaftor; deutivacaftor, tezacaftor , vanzacaftor

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- Part A: Single Ascending Dose (SAD) (Experimental): Participants will be randomized to receive a single dose of different dose levels of VX-828.
  Interventions: Drug: VX-828
- Part A: Placebo (Placebo Comparator): Participants will be randomized to receive placebo matched to VX-828.
  Interventions: Drug: Placebo
- Part B: Multiple Ascending Dose (MAD) (Experimental): Participants will be randomized to receive multiple doses of different dose levels of VX-828. The dose levels will be determined based on the data from Part A.
  Interventions: Drug: VX-828
- Part B: Placebo (Placebo Comparator): Participants will be randomized to receive placebo matched to VX-828.
  Interventions: Drug: Placebo
- Part C: Drug Drug Interaction (Experimental): Participants will receive a single dose of VX-828, followed by a washout period, Itraconazole administration, and concomitant administration of itraconazole and VX-828; or participants will receive Midazolam followed by VX-828/TEZ/D-IVA administration, and concomitant administration of VX-828/TEZ/D-IVA and Midazolam.
  Part C will be an open-label optional cohort.
  Interventions: Drug: VX-828; Drug: Itraconazole; Drug: Midazolam; Drug: Tezacaftor; Drug: Deutivacaftor
- Part D: VX-828 in combination with TEZ/VX-118 ,TEZ/D-IVA or D-IVA (Experimental): Participants will be randomized to receive VX-828 in combination with TEZ/VX-118, TEZ/D-IVA, or D-IVA.
  Interventions: Drug: VX-828; Drug: Tezacaftor; Drug: VX-118; Drug: Deutivacaftor
- Part D: Placebo (Placebo Comparator): Participants will be randomized to receive placebo matched to VX-828/TEZ/VX-118 or placebo matched to VX-828 in combination with TEZ/D-IVA or D-IVA
  Interventions: Drug: Tezacaftor; Drug: Placebo; Drug: Deutivacaftor
- Part E: VX-828 in Combination with D-IVA with or without TEZ in CF (Experimental): Participants with cystic fibrosis will receive VX-828 in combination with D-IVA with or without TEZ.
  Interventions: Drug: Tezacaftor; Drug: Deutivacaftor; Drug: VX-828

INTERVENTIONS:
Drug: VX-828 — Suspension for Oral Administration
  Arms: Part A: Single Ascending Dose (SAD); Part B: Multiple Ascending Dose (MAD); Part C: Drug Drug Interaction; Part D: VX-828 in combination with TEZ/VX-118 ,TEZ/D-IVA or D-IVA
Drug: Placebo — Suspension for Oral Administration
  Arms: Part A: Placebo; Part B: Placebo
Drug: Itraconazole — Solution for Oral Administration
  Arms: Part C: Drug Drug Interaction
Drug: Midazolam — Syrup for Oral Administration
  Arms: Part C: Drug Drug Interaction
Drug: Tezacaftor — Tablets for Oral Administration
  Other Names: TEZ; VX-661
  Arms: Part C: Drug Drug Interaction; Part D: Placebo; Part D: VX-828 in combination with TEZ/VX-118 ,TEZ/D-IVA or D-IVA; Part E: VX-828 in Combination with D-IVA with or without TEZ in CF
Drug: VX-118 — Tablets for Oral Administration
  Arms: Part D: VX-828 in combination with TEZ/VX-118 ,TEZ/D-IVA or D-IVA
Drug: Placebo — Suspension and Tablets for Oral Administration
  Arms: Part D: Placebo
Drug: Deutivacaftor — Tablets for Oral Administration
  Other Names: D-IVA; VX-561
  Arms: Part C: Drug Drug Interaction; Part D: Placebo; Part D: VX-828 in combination with TEZ/VX-118 ,TEZ/D-IVA or D-IVA; Part E: VX-828 in Combination with D-IVA with or without TEZ in CF
Drug: VX-828 — Tablets for Oral Administration
  Arms: Part E: VX-828 in Combination with D-IVA with or without TEZ in CF

SUMMARY:
The purpose of the study is to evaluate safety, tolerability, and pharmacokinetics of VX-828 and VX-828 in triple combination (TC) with Tezacaftor (TEZ)/ VX-118 or TEZ/ deutivacaftor (D-IVA) in healthy participants and VX-828 in combination with D-IVA with or without TEZ in participants with cystic fibrosis (CF).

DETAILED DESCRIPTION:
This clinical trial information was submitted voluntarily under the applicable law and, therefore, certain submission deadlines may not apply. (That is, clinical trial information for this applicable clinical trial was submitted under section 402(j)(4)(A) of the Public Health Service Act and 42 CFR 11.60 and is not subject to the deadlines established by sections 402(j)(2) and (3) of the Public Health Service Act or 42 CFR 11.24 and 11.44.).

ELIGIBILITY:
Key Inclusion Criteria:

Parts A-D:

* Participants between the ages of 18 and 55 years
* Body mass index (BMI) of 18.0 to 32.0 kilogram per meter square (kg/m^2)
* A total body weight of more than (>) 50 kg
* Nonsmoker or ex-smoker for at least 3 months before screening with current nonsmoking status confirmed by urine or blood cotinine at screening
* Cohort C2 only: Willing to provide a single DNA sample

Part E:

* Participants 18 years or older
* Confirmed diagnosis of CF as determined by the investigator
* A total body weight of more than or equal to (>=) 35 kg
* Participants must be heterozygous for F508del with a second CFTR allele carrying a minimal function mutation that is not responsive to ELX/TEZ/IVA therapy
* Participants must have a forced expiratory volume in 1 second (FEV1) of greater than or equal to (≥) 40% of predicted normal for age, sex, and height

Key Exclusion Criteria:

Parts A-D:

* History of febrile illness or other acute illness within 14 days before the first dose of study drug
* Any condition possibly affecting drug absorption

Part E:

* An acute illness not related to CF (e.g., gastroenteritis) within 14 days before the first dose of study drug
* History of solid organ or hematological transplantation
* History of clinically significant cirrhosis with or without portal hypertension
* Lung infection with organisms associated with a more rapid decline in pulmonary status

Other protocol defined Inclusion/Exclusion criteria will apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 255 (Estimated)
Dates: Start 2023-12-12 (Actual); Primary Completion 2026-04-23 (Estimated); Study Completion 2026-04-23 (Estimated)

PRIMARY OUTCOMES:
Part A: Safety and Tolerability as Assessed by Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs) | From Signing of Informed Consent Form (ICF) up to Safety Follow Up (Up to Day 67)
Part B: Safety and Tolerability as Assessed by Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs) | From Signing of Informed Consent Form (ICF) up to Safety Follow Up (Up to Day 80)
Part D: Safety and Tolerability as Assessed by Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs) | From Signing of Informed Consent Form (ICF) up to Safety Follow Up (Up to Day 80)
Part E: Safety and Tolerability as Assessed by Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs) | From Signing of Informed Consent Form (ICF) up to End of Study (Up to Day 111)
Part C: Maximum Observed Concentration (Cmax) of VX-828 in Plasma in the Absence and Presence of Itraconazole | From Day 1 up to Day 71
Part C: Area Under the Concentration Versus Time Curve (AUC) of VX-828 in Plasma in the Absence and Presence of Itraconazole | From Day 1 up to Day 71
Part C: Maximum Observed Concentration (Cmax) of Midazolam in Plasma in the Absence and Presence of VX-828/TEZ/D-IVA | From Day 1 up to Day 30
Part C: Area Under the Concentration Versus Time Curve (AUC) of Midazolam in Plasma in the Absence and Presence of VX-828/TEZ/D-IVA | From Day 1 up to Day 30

SECONDARY OUTCOMES:
Part A: Maximum Observed Concentration (Cmax) of VX-828 in Plasma | From Day 1 up to Day 67
Part A: Area Under the Concentration Versus Time Curve (AUC) of VX-828 in Plasma | From Day 1 up to Day 67
Part B: Maximum Observed Concentration (Cmax) of VX-828 at Day 28 in Plasma | From Day 1 up to Day 80
Part B: Area Under the Concentration Versus Time Curve (AUC) of VX-828 at Day 28 in Plasma | From Day 1 up to Day 80
Part C: Safety and Tolerability as Assessed by Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs) | From Signing of Informed Consent Form (ICF) up to Safety Follow Up (Up to Day 82)
Part D: Maximum Observed Concentration (Cmax) of VX-828, TEZ and D-IVA and their Metabolites at Day 28 in Plasma | Day 28
Part D: Area Under the Concentration Versus Time Curve (AUC) of VX-828, TEZ and D-IVA and their Metabolites at Day 28 in Plasma | Day 28
Part E: Maximum Observed Concentration (Cmax) of VX-828, TEZ, and D-IVA and their Metabolites in Plasma | Day 1 and Day 28
Part E: Area Under the Concentration Versus Time Curve (AUC) of VX-828, TEZ, and D-IVA and their Metabolites in Plasma | Day 28
Part E: Pre-dose Plasma Concentration (Ctrough) of VX-828, TEZ, D-IVA and its Metabolites | Pre-dose at Day 4, Day 8, Day 15, Day 22, Day 35, Day 49, Day 63, Day 80
Part E: Absolute Change in Sweat Chloride | From Baseline and At Day 28

CONTACTS AND LOCATIONS:
Locations (11):
- United States (11):
  - Joe DiMaggio Cycstic Fibrosis & Pulmonary Center, Hollywood, Florida
  - Central Florida Pulmonary Group, P.A., Orlando, Florida
  - Altasciences Clinical Kansas, Overland Park, Kansas
  - Kentucky Children's Hospital, Lexington, Kentucky
  - Boston Children's Hospital, Boston, Massachusetts
  - University of Minnesota -Pulmonology, Minneapolis, Minnesota
  - New York Medical College, Hawthorne, New York
  - ProMedica Toledo Children's Hospital & ProMedica Central Physicians, LLC, Toledo, Ohio
  - Cook Children's Pulmonology, Fort Worth, Texas
  - University of Utah Hospital - Pulmonology, Salt Lake City, Utah
  - Vermont Lung Center, Colchester, Vermont

IPD SHARING:
Plan to Share IPD: No
Details on Vertex data sharing criteria and process for requesting access can be found at: https://www.vrtx.com/our-science/clinical-trials-data-sharing/